CLINICAL TRIAL: NCT04312880
Title: Tranexamic Acid Infusion During Elective Spine Surgery
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5176
Record Dates: First submitted 2020-03-09; First posted 2020-03-18 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Spine Surgery
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Patient will receive no transexemic acid of any kind
- IV-transexemic acid (Experimental): weight adjusted standard dose of TXA will be administered to these subset of patients prior to incision in IV-form
  Interventions: Drug: Tranexamic Acid
- Topical-transexemic acid (Experimental): the wound site after the surgery is completed will be bathed in TXA for a standardized period of time prior to skin closure
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — IV and topical form of TXA will be administered to patients in the respective groups.
  Arms: IV-transexemic acid; Topical-transexemic acid

SUMMARY:
Tranexamic acid (TXA) is an agent that has been shown to be safe and effective to reduce blood loss in surgical procedures. The purpose of the study is to assess the effect of transexamic on elective decompressive lumbar spine surgery with and without fusion.

DETAILED DESCRIPTION:
This will be a prospective randomized control, double-blinded investigation. The Investigators will recruit patients undergoing elective, primary, decompressive lumbar surgery via a posterior surgical approach of less than 3 levels. This includes patients undergoing decompressive lumbar laminectomies with or without fusion. Fusion may include posterior interbody and/or posterior lateral techniques with instrumentation.

There will be 3 treatment arms with the goal of 65 patients in each arm. Patients will be randomized pre-operatively and enrolled into the IV transexamic acid group (receiving intraoperative intravenous tranexamic acid infusion), or the topical transexamic acid group or the control/placebo group (receiving intraoperative intravenous saline). The Investigators expect the duration of each treatment group to be approximately 4-5 months. Therefore, the study should be completed within 1.5 years. The primary surgeon and anesthesia staff will not be blinded to the treatment arm due to the nature of the different administration routes, but post-operative nursing staff will be blinded to administration routes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing decompressive lumbar laminectomy with or without fusion
* Primary surgical procedure
* Competent adult able to give informed consent
* Age >18

Exclusion Criteria:

* h/o DVT or PE
* h/o seizure
* h/o coagulopathy
* Diagnosis of malignancy or infection as indication for surgical decompression
* Abnormal pre-operative PT/INR, aPTT, bleeding time
* Platelet count < 100
* Patients requiring therapeutic heparin or lovenox bridges prior to and/or after surgery
* Allergy to TXA
* Pregnant women and prisoners
* Renal insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Drain output | 48 hours postoperatively
  Drains will be placed during surgery, this will be recorded by nursing staff on a regular schedule and we will assess the results as a surrogate for blood loss post operatively

SECONDARY OUTCOMES:
Change in hematocrit | two days post operatively
  Labs will be recorded each morning after the surgery, this includes hematocrit
Change in hemoglobin | two days post operatively
  Labs will be recorded each morning after the surgery, this includes hemoglobin
Emergency department visits | 30 days post operatively
  We will assess which treatment arms, if any had increased rate of Emergency department visits for any reason
number of hospital readmissions | 30 days post operatively
  We will assess which treatment arms, if any had increased rate of readmission to the hospital
Incidence of PE | 30 days post opertively
  We will assess is any treatment arm had an increased risk of PE
Incidence of DVT | 30 days post opertively
  We will assess is any treatment arm had an increased risk of DVT

CONTACTS AND LOCATIONS:
Overall Officials: James Lawrence, MD, Principal Investigator — Attending Surgeon
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No